CLINICAL TRIAL: NCT06464848
Title: Narrative Identity and Its Relationship to Subjective Multidimensional Well-being in First Episode Psychosis
Acronym: PEPsy-Identity
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2023/JJ-03
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Psychosis
Keywords: First episode psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- FEP: Participants recruited from PEPsy-CM trial
  Interventions: Other: Narrative identity task
- Chronic: Participants recruited from psychiatric department of CHU de Nimes
  Interventions: Other: Narrative identity task
- Controls: Recruited from social media and word of mouth
  Interventions: Other: Narrative identity task

INTERVENTIONS:
Other: Narrative identity task — All participants will be asked to develop five personal narratives in response to different types of questions: trauma, transgression, negative memory, self-definition, and turning point. For each story, participants will be asked to provide details of where they were, who they were with, what happened and how they and others reacted, what happened, how they reacted and how others reacted (if at all).

SUMMARY:
The transition between adolescence and adulthood (generally defined as ages 18 to 25) is a key developmental window for narrative identity and psychotic disorders. Narrative identity is positively associated with mental health. This study will focus on the acquisition of narrative identity in First Episode Psychosis (FEP) and its impact on multidimensional subjective well-being.

The study authors hypothesize that levels of the various components of narrative identity would be lower in the FEP group than in the "chronic" and control groups, and in the "chronic" group versus control group. Given the paucity contradictory nature of the published literature, no hypotheses have been formulated regarding these correlations and predictions. Instead, this study will remain an exploratory analysis in the different samples.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Inclusion criteria fir FEP group:

• Patient managed in the psychiatry department (consultation or hospitalization) for a FEP defined by :

* Presence of positive psychotic symptoms (delirium(s) and/or hallucination(s) and/or conceptual disorganization) for at least one week, either every day or at least 3 times a week for at least one hour.
* Never having taken neuroleptic antipsychotic treatment (except antipsychotic treatment started for the current episode)
* Disorder meeting DSM 5 criteria from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific disorder of the schizophrenic spectrum or other psychotic disorder, bipolar I or II disorder with psychotic features congruent and not congruent with mood, substance-induced bipolar disorder with psychotic features congruent and not congruent with mood, major depressive disorder with psychotic features congruent and not congruent with mood.

Inclusion criteria for the "Chronic" group:

• Patient diagnosed with a disorder meeting DSM 5 criteria for more than 18 months from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific disorder of the schizophrenic spectrum or other psychotic disorder, bipolar I or II disorder with psychotic features congruent and not congruent with mood, substance-induced bipolar disorder with psychotic features congruent and not congruent with mood, major depressive disorder with psychotic features congruent and not congruent with mood.

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject unable to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient pregnant or breastfeeding
* Patient with history of traumatic brain injury
* Patient with moderate to severe mental retardation (IQ≤ 55)

Exclusion criteria for FEP group:

• FEP related to a drug-induced psychotic disorder or due to another medical condition

Exclusion criteria for the "Control" group:

* Participant with lifetime experience of FEP
* Participant with a diagnosis of a disorder meeting DSM 5 criteria from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific disorder of the schizophrenic spectrum or other psychotic disorder, bipolar I or II disorder with psychotic features congruent and not congruent with mood, substance-induced bipolar disorder with psychotic features congruent and not congruent with mood, major depressive disorder with psychotic features congruent and not congruent with mood.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of three study groups:
  1. Patients with a first psychotic episode (FEP group)
  2. Controls, representative of the general French population (control group)
  3. Patients with a diagnosis of psychotic or bipolar disorder ("chronic" group). All three groups will be matched for age, sex and socio-educational level.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Narrative identity between groups according to life history task | Day 0
  Narrative identity calculated from five narratives scored by the clinician considering agency, communion, redemption/contamination, affective tone, exploratory processing, growth, construction of meaning, elaboration of facts and interpretations, affective tone, ending valence, temporal/causal/thematic coherence and overall coherence.

SECONDARY OUTCOMES:
Multidimensional subjective well-being between groups | Day 0
  PERMA-Profiler score. A 15-item questionnaire measured on 11-item Likert scales. Higher scores indicate greater well-being. An overall well-being score is calculated by creating an average score for each item, and subscale scores are calculated by averaging the three items in each subscale
Psychopathology symptoms between FEP and chronic groups | Day 0
  Positive and negative symptom scale (PANSS). The positive scale ranges from 7 to 49, the negative scale from 8 to 56, the hostility scale from 6 to 46, the disorganization scale from 5 to 35, and the anxiety scale from 4 to 28. The total score ranges from 30 to 210.
Personal recovery between FEP and chronic groups | Day 0
  Stage of Recovery Instrument (STORI). Ten themes are evaluated, each comprising five items ranging from 0 "Not at all true" to 5 "Quite true", corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50, and the participant is assigned to the stage with the highest score.
Personality between groups | Day 0
  10-item Big Five Inventory (BFI-10). The BFI-10 is a 10-item scale assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability and openness
Childhood trauma between groups | Day 0
  Childhood Trauma Questionnaire (CTQ). The short version of the CTQ consists of 28 items, including a 3-item denial scale and five 5-item scales. The scale items are a Likert-type scale with five response options (from 1 = "never true" to 5 = "very often true")
Patient functioning between groups | Day 0
  Global Assessment of Functioning (GAF). Scores range from 0-100, whereby lower scores represent lower functioning
Anxiety and depression between groups | Day 0
  Hospital Anxiety and Depression Scale (HADS). A 14-item questionnaire of which 7 assess depression and 7 anxiety. The sum of the item scores for each subscale produces an anxiety score and/or a depression score
Social and individual performance between groups | Day 0
  Personal and Social Performance scale (PSP). Higher scores correspond to better personal and social functioning, scores from 91 to 100 correspond to more than adequate functioning, while scores below 30 correspond to such poor functioning that intensive supervision is required
General quality of life between groups | Day 0
  World Health Organization Quality Of Life Brief (WHOQOL-BREF). The WHOQOL-bref has four types of five-point response scales, allowing assessment of intensity (Not at all-Extremely), ability (Not at all-Completely), frequency (Never-Always) and evaluation (Very dissatisfied/Very bad-Very satisfied/Very good), which vary according to the items
Autobiographical memory function between groups | Day 0
  Thinking About Life Experiences scale (TALE-15). This self-questionnaire consists of two general questions, followed by 15 items specific to autobiographical memory functions, each consisting of 5 items. The response items are associated with a 5-point Likert scale ranging from "Almost never" to "Very frequently".
Insight between FEP and chronic groups | Day 0
  Birchwood Insight Scale (BIS). The questionnaire measures multidimensional assessment of insight, comprising 8 questions (3-point Likert scale: "agree", "disagree" or "unsure"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Health-related quality of life between groups | Day 0
  EuroQol-5Dimension (EQ-5D-5L) questionnaire. This questionnaire comprises five items representing the 5 dimensions of quality of life and a 0-100 visual analog scale. The answers are combined into a 5-digit number describing the patient's health status e.g., health status "11111" indicates the absence of problems
Depression between groups | Day 0
  Beck Depression Inventory (BDI-11).
Medical adherence between FEP and chronic groups | Day 0
  Medication Adherence Rating Scale (MARS). The 10 items assess behaviors, attitudes and treatment experience. Scores range from 0 to 10
Patient-perceived improvement in clinical condition between FEP and chronic groups | Day 0
  Clinical Global Impression (CGI). The questionnaire comprises two measures: Severity and Improvement, both measured on a scale of 1 to 7
Verbal fluency between groups | Day 0
  Participants must list as many words as possible beginning with the letter "P", belonging to the semantic category "animals".
Word recall and recognition between groups | Day 0
  California Verbal Learning Test (CVLT-11). Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall). The word list is presented as a shopping list.
Non-verbal reasoning between groups | Day 0
  Matrices test taken from the Wechsler Adult Intelligence Scale to measure non-verbal reasoning abilities, general visual intelligence and perceptual organization skills.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Jourdan, Principal Investigator — CHU de Nimes
Locations (1):
- Department of Psychiatry, Nimes University Hospital, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No